CLINICAL TRIAL: NCT05867524
Title: Characterization of Natural IL-6 Inhibition in Healthy Individuals
Acronym: FIDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Clinical Immunological Department, Rigshospitalet (Unknown); The Danish Blood Donor Study (Unknown)
Responsible Party: Principal Investigator, Torben Hansen, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-20082776
Record Dates: First submitted 2023-01-27; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Autoantibodies; Interleukin-6
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Groups defined by autoantibodies status (high or low)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High IL-6 c-aAb (Experimental): Individuals with top percentile IL-6 c-aAb
  Interventions: Other: Oral Glucose Tolerance Test; Other: Cycling test
- Low IL-6 c-aAb (Experimental): Individually matched controls with low IL-6 c-aAb
  Interventions: Other: Oral Glucose Tolerance Test; Other: Cycling test

INTERVENTIONS:
Other: Oral Glucose Tolerance Test — 75g oral glucose tolerance test, sampled over three hours
Other: Cycling test — 2 hours of moderate activity level cycling

SUMMARY:
The aim of the project is to investigate whether or not there are any difference in cardiometabolic outcomes in individuals with high or low levels of c-aAb against interleukin-6 (IL-6).

The study is the first to investigate individuals with extreme amounts of c-aAb levels against IL-6 and to contribute with knowledge on a possible new phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill Danish blood donor criteria
* Have extreme amounts of IL-6 c-aAb or matched as control (low amounts of IL-6 c-aAb)

Exclusion Criteria:

* Failure to fulfill Danish blood donor criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  IL-6 plasma levels, plasma IL-6 c-aAb levels
Whole-body glucose metabolism | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Plasma levels of: Insulin
Whole-body glucose metabolism | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Plasma levels of: C-peptide
Whole-body glucose metabolism | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Plasma levels of: Glucose
Whole-body glucose metabolism | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Plasma levels of: GLP-1
Whole-body glucose metabolism | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Plasma levels of: GIPR
Cardiovascular risk markers | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Lipids
Cardiovascular risk markers | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Triglyceride
Cardiovascular risk markers | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Blood pressure
Cardiovascular risk markers | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Epicardial adipose tissue
Difference in exercise response | Measurements over a two-hour cycling test, and one hour of recovery
  2-hour Lactate
Difference in exercise response | Measurements over a two-hour cycling test, and one hour of recovery
  2-hour epinephrine
Difference in exercise response | Measurements over a two-hour cycling test, and one hour of recovery
  2-hour norepinephrine
Difference in exercise response | Measurements over a two-hour cycling test, and one hour of recovery
  Peak IL-6
Metabolic response during exercise | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  2-hour glucose
Metabolic response during exercise | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  2-hour glucagon
Metabolic response during exercise | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  2-hour insulin
Metabolic response during exercise | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  2-hour lipids
Metabolic response during exercise | Measurements over a three-hour oral glucose tolerance test, a two-hour cycling test, and one hour of recovery
  Triglyceride
Metabolic assessment of the liver | An MRI-scanning withinn four weeks of the oral glucose tolerance test
  Liver fat content from MRI-scanning, and HOMA-IR
Metabolic assessment of the liver | An MRI-scanning withinn four weeks of the oral glucose tolerance test
  HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Torben Hansen, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No